CLINICAL TRIAL: NCT04925765
Title: Virtual Reality Biofeedback for Postpartum Anxiety and Depression
Acronym: VITALISE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Grace Lim, MD, MS (Other)
Responsible Party: Sponsor-Investigator, Grace Lim, MD, MS, Associate Professor, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY21040063
Record Dates: First submitted 2021-06-07; First posted 2021-06-14 (Actual); Results first posted 2024-04-17 (Actual); Last update posted 2024-04-17 (Actual); Status verified 2024-04

CONDITIONS: Anxiety and Depression; Postpartum Depression; Pregnancy Related
MeSH Terms: conditions — Anxiety Disorders; Depression; Depression, Postpartum

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Virtual Reality (VR) Session (Experimental): All participants in this study will complete a 1 hour virtual reality session.
  Interventions: Other: Virtual Reality Biofeedback Session

INTERVENTIONS:
Other: Virtual Reality Biofeedback Session — The "Flowly" intervention treatment utilizes virtual reality and biofeedback to train patients to auto-regulate themselves and improve their pain/anxiety/depression.

SUMMARY:
The purpose of this study is to test patient feasibility and acceptability of virtual reality biofeedback program in postpartum women for anxiety and depression outcomes.

DETAILED DESCRIPTION:
In an open-label pilot trial, women will undergo a single session using the virtual reality biofeedback program. The objective of this study is to assess feasibility and acceptability of virtual reality biofeedback program in postpartum women with specific assessments of anxiety and depression outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Currently pregnant or postpartum (delivery within 3 months)
* 18 years or older

Exclusion Criteria:

* Unable to participate in study procedures
* English illiterate (surveys validated in English)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2021-09-30 (Actual); Study Completion 2021-10-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Grace Lim, MD,MS, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Stamou G, Garcia-Palacios A, Botella C. Cognitive-Behavioural therapy and interpersonal psychotherapy for the treatment of post-natal depression: a narrative review. BMC Psychol. 2018 Jun 18;6(1):28. doi: 10.1186/s40359-018-0240-5. PMID 29914574
- [Background] Kolbe L, Jaywant A, Gupta A, Vanderlind WM, Jabbour G. Use of virtual reality in the inpatient rehabilitation of COVID-19 patients. Gen Hosp Psychiatry. 2021 Jul-Aug;71:76-81. doi: 10.1016/j.genhosppsych.2021.04.008. Epub 2021 Apr 29. PMID 33964789
- [Background] Baschong A, Spiess F, Cattin PC, Navarini A, Mueller SM. Itch reduction using immersive virtual reality-An experimental pilot study. Dermatol Ther. 2021 Jul;34(4):e15001. doi: 10.1111/dth.15001. Epub 2021 Jun 9. PMID 34036696
- [Background] Vlake JH, Van Bommel J, Wils EJ, Korevaar TIM, Hellemons ME, Schut AFC, Labout JAM, Schreuder LLH, Gommers D, Van Genderen ME. Effect of intensive care unit-specific virtual reality (ICU-VR) to improve psychological well-being and quality of life in COVID-19 ICU survivors: a study protocol for a multicentre, randomized controlled trial. Trials. 2021 May 5;22(1):328. doi: 10.1186/s13063-021-05271-z. PMID 33952318
- [Background] Sasseville M, LeBlanc A, Boucher M, Dugas M, Mbemba G, Tchuente J, Chouinard MC, Beaulieu M, Beaudet N, Skidmore B, Cholette P, Aspiros C, Larouche A, Chabot G, Gagnon MP. Digital health interventions for the management of mental health in people with chronic diseases: a rapid review. BMJ Open. 2021 Apr 5;11(4):e044437. doi: 10.1136/bmjopen-2020-044437. PMID 33820786
- [Background] Alneyadi M, Drissi N, Almeqbaali M, Ouhbi S. Biofeedback-Based Connected Mental Health Interventions for Anxiety: Systematic Literature Review. JMIR Mhealth Uhealth. 2021 Apr 22;9(4):e26038. doi: 10.2196/26038. PMID 33792548
- [Background] Polat M, Kahveci A, Muci B, Gunendi Z, Kaymak Karatas G. The Effect of Virtual Reality Exercises on Pain, Functionality, Cardiopulmonary Capacity, and Quality of Life in Fibromyalgia Syndrome: A Randomized Controlled Study. Games Health J. 2021 Jun;10(3):165-173. doi: 10.1089/g4h.2020.0162. Epub 2021 Mar 9. PMID 33689452
- [Background] Turrado V, Guzman Y, Jimenez-Lillo J, Villegas E, de Lacy FB, Blanch J, Balibrea JM, Lacy A. Exposure to virtual reality as a tool to reduce peri-operative anxiety in patients undergoing colorectal cancer surgery: a single-center prospective randomized clinical trial. Surg Endosc. 2021 Jul;35(7):4042-4047. doi: 10.1007/s00464-021-08407-z. Epub 2021 Mar 8. PMID 33683433

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Postpartum women with a history of anxiety (ANX) or depression (DEP) participated in a single virtual reality (VR) biofeedback session.
Pre-assignment Details: All women who were willing to participate received the same treatment arm, VR biofeedback session.
Groups:
- Virtual Reality Session: All participants in this study will complete a 1 hour virtual reality session.
  Flowly (TMC-CP01): The Flowly (TMC-CP01) treatment utilizes virtual reality and biofeedback to train patients to auto-regulate themselves and improve their pain/anxiety/depression.
Period: Overall Study
Arm/Group | Virtual Reality Session
Started | 6
Completed | 6
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Virtual Reality Session
Number analyzed (Participants) | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 6
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.9 (4.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: number of participants]
  United States | 6
Anxiety [Mean (Standard Deviation); unit: units on a scale] — Measure of participant's baseline state and trait anxiety. Consists of 40 questions based on a 4-point Likert scale. High scores are positively correlated with high levels of anxiety. Scores range from 0-120.
  units on a scale | 42.3 (10.3)
Depression at baseline [Mean (Standard Deviation); unit: units on a scale] — Baseline depression measured via Edinburgh Postnatal Depression Scale, a 10-item questionnaire with a minimum score of 0 and a maximum score of 30. A score of 10 or greater is indicative of possible depression, a score of 14 or greater is indicative of severe depression.
  units on a scale | 6.3 (3.5)

OUTCOME MEASURES:

1. Primary Outcome: Intervention Feasibility
Description: Patient response to the feasibility of VR use. The question asked was, "I was able to do the session without difficulty," which was measured on a Likert Scale of 1-5. A score of 1 is indicative of great difficulty present and a score of 5 is indicative of no difficulty present. Outcome measurement is presented as an averaged score with standard deviation among participating patients.
Time Frame: Completed immediately after the VR session.
Population: postpartum women
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Virtual Reality Session
Number analyzed (Participants) | 6
score on a scale | 4.83 (0.41)

2. Primary Outcome: Intervention Acceptability
Description: Acceptability was assessed by questions, "Would you participate in another session?" Acceptability was measured by yes/no responses and reported as an overall percentage of participating patients who responded as yes.
Time Frame: Completed directly after the VR intervention session and anxiety/depression measurements.
Population: postpartum women
Measure: Count of Participants; unit: Participants
Arm/Group | Virtual Reality Session
Number analyzed (Participants) | 6
Participants | 5

3. Secondary Outcome: Decrease in Depression From Baseline to Post-intervention
Description: Number of participants whose depression scores (as measured by Edinburgh Postnatal depression scale (EPDS)) decreased from baseline to post-VR intervention.
Time Frame: EPDS Completed directly before and after VR session.
Population: number of participants whose depression scores decreased.
Measure: Count of Participants; unit: Participants
Arm/Group | Virtual Reality Session
Number analyzed (Participants) | 6
Participants | 5

4. Secondary Outcome: Decrease in State-Trait Anxiety Inventory (STAI) From Baseline to Post-intervention
Description: Number of participants whose anxiety scores (as measured by STAI) decreased from baseline to post-VR intervention.
Time Frame: Completed directly before and after VR session.
Population: Number of participants with decreases in anxiety scores pre-post.
Measure: Count of Participants; unit: Participants
Arm/Group | Virtual Reality Session
Number analyzed (Participants) | 6
Participants | 5

ADVERSE EVENTS:
Time Frame: Within the study intervention of 2 hours.
Arm/Group | Virtual Reality Session
All-Cause Mortality (participants affected / at risk) | 0/6
Serious Adverse Events (participants affected / at risk) | 0/6
Other Adverse Events (participants affected / at risk) | 0/6

LIMITATIONS AND CAVEATS:
The study is limited by the exploratory nature and small sample size, but feasibility is appropriate to assess in a clinical setting.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-09-05): https://cdn.clinicaltrials.gov/large-docs/65/NCT04925765/Prot_SAP_000.pdf